CLINICAL TRIAL: NCT01365624
Title: A Phase 1 Safety and Pharmacokinetics Study of Intranasal Ketorolac in Elderly and Nonelderly Adult Healthy Subjects
Brief Title: Safety and Pharmacokinetics Study of Intranasal Ketorolac in Elderly and Nonelderly Adult Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: American Regent, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ROX 2007-02
Record Dates: First submitted 2011-06-01; First posted 2011-06-03 (Estimated); Results first posted 2013-02-06 (Estimated); Last update posted 2013-02-06 (Estimated); Status verified 2013-01

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — Ketorolac Tromethamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ketorolac tromethamine (Experimental)
  Interventions: Drug: Ketorolac tromethamine

INTERVENTIONS:
Drug: Ketorolac tromethamine — Single dose of 30 mg of intranasal Ketorolac tromethamine (100 uL of a 15% solution in each nostril)

SUMMARY:
This study had an open-label, single-dose design. All subjects received a single dose of 30 mg of intranasal ketorolac. Blood samples for determination of ketorolac plasma levels were obtained pre-dose and at specified time points over 24 hours post-dose.

The primary objective of this trial was to compare the pharmacokinetics of intranasal ketorolac between elderly and nonelderly adult subjects. The secondary objective was to evaluate the safety profile of intranasal ketorolac in elderly subjects.

ELIGIBILITY:
Inclusion Criteria:

* The elderly population consisted of male or female volunteers aged > of = 65 years
* The nonelderly adult population consisted of male or female volunteers aged < 65 years
* Generally good health in the opinion of the Investigator, as determined by a prestudy physical examination with no clinically significant abnormalities for age, vital signs within normal ranges or outside normal range but not deemed clinically significant for age in the opinion of the Investigator, and no clinically significant electrocardiogram (ECG) abnormalities for age
* Bilaterally patent nasal airways at screening as assessed by the Investigator
* Body mass index (BMI) 15-30 kg/m2
* Female subjects of childbearing potential must consent to use a medically acceptable method of contraception (oral or implanted contraceptive hormones, condom or diaphragm with spermicidal agent, intrauterine device, or surgical sterilization) throughout the study period
* Ability to provide written informed consent
* Prestudy clinical laboratory findings within normal ranges or if outside normal range not deemed clinically significant for age in the opinion of the Investigator

Exclusion Criteria:

* Allergy or sensitivity to ketorolac or formulation ingredients
* History of co-existing nasal polyps, NSAID sensitivity, and asthma
* Allergic reaction to aspirin or other NSAIDs
* Current upper respiratory tract infection or other respiratory tract condition that could interfere with the absorption of the nasal spray or with the assessment of AEs
* Use of any prescribed or over-the-counter (OTC) drug in the 72 h prior to entry into the study with the exception of occasional acetaminophen up to 24 h prior to entry
* Suspicion of rhinitis medicamentosa (chronic daily use of topical decongestants)
* Use of a monoamine oxidase (MAO) inhibitor in the 14 days prior to study entry
* Positive serum test for human immunodeficiency virus (HIV) or hepatitis B or C
* Positive alcohol breath test at screening or on entry into the study
* Positive urine screen for any nonprescribed drug of abuse at screening or on entry into the study
* History of cocaine use
* Blood donation within 30 days of beginning study participation
* Active peptic ulcer disease or a history of peptic ulcer disease or gastrointestinal bleeding
* Serum creatinine > 2.0 mg/dL
* Current tobacco use or a past history of smoking within 5 years of study entry
* Any other clinically significant medical problem, which in the opinion of the Investigator would interfere with study participation
* Participation within 30 days of study entry or within 5 times the half-life, whichever is longer, in another investigational drug study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-02; Primary Completion 2008-04 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lincoln Bynum, MD, Study Chair — ICON Developmental Solutions
Locations (1):
- Seaview Research, Miami, Florida, United States

REFERENCES:
- [Derived] Bullingham R, Juan A. Comparison of intranasal ketorolac tromethamine pharmacokinetics in younger and older adults. Drugs Aging. 2012 Nov;29(11):899-904. doi: 10.1007/s40266-012-0023-2. PMID 23143939

RESULTS

PARTICIPANT FLOW:
Recruitment Details: February 2008 through April 2008; Clinical Unit
Pre-assignment Details: After subjects had given their informed consent, subjects were required to pass a screening visit within 3 weeks prior to study drug administration.
Groups:
- Ketorolac Tromethamine (Elderly Adults ≥ 65); Ketorolac Tromethamine (Nonelderly Adults < 65): Ketorolac tromethamine : Single dose of 30 mg of intranasal Ketorolac tromethamine (100 uL of a 15% solution in each nostril)
Period: Overall Study
Arm/Group | Ketorolac Tromethamine (Elderly Adults ≥ 65) | Ketorolac Tromethamine (Nonelderly Adults < 65)
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ketorolac Tromethamine (Elderly Adults ≥ 65) | Ketorolac Tromethamine (Nonelderly Adults < 65) | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 15 | 15
  >=65 years | 15 | 0 | 15
Age Continuous [Mean (Standard Deviation); unit: years] | 71.9 (5.9) | 44.2 (10.3) | 58.1 (16.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 14
  Male | 7 | 9 | 16
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Cmax (Maximum Plasma Concentration)
Time Frame: Blood samples for PK analyses were obtained at pre-dose (15 minutes prior to ketorolac administration), 15 minutes, 30 minutes, 45 minutes, 1 hour, 1 hour and 30 minutes, 2 hours, 4 hours, 6 hours, 8 hours, 12 hours, 15 hours and 24 hours post-dose
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Ketorolac Tromethamine (Elderly Adults ≥ 65) | Ketorolac Tromethamine (Nonelderly Adults < 65)
Number analyzed (Participants) | 15 | 15
ng/mL | 1782.286 (1184.843) | 1840.111 (995.930)

2. Primary Outcome: Tmax (Time to Reach Maximum Plasma Concentration)
Time Frame: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Ketorolac Tromethamine (Elderly Adults ≥ 65) | Ketorolac Tromethamine (Nonelderly Adults < 65)
Number analyzed (Participants) | 15 | 15
hours | 0.750 [0.50 to 1.00] | 0.750 [0.25 to 1.00]

3. Primary Outcome: AUClast (Area Under the Plasma Concentration-time Profile From Time Zero to the Last Quantifiable Time Point Post-dose
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*hours/mL
Arm/Group | Ketorolac Tromethamine (Elderly Adults ≥ 65) | Ketorolac Tromethamine (Nonelderly Adults < 65)
Number analyzed (Participants) | 15 | 15
ng*hours/mL | 7323.5 (4633.1) | 6536.5 (3361.8)

4. Primary Outcome: AUC (Area Under the Plasma Concentration-time Profile From Time 0 to Infinity
Time Frame: as for outcome 1
Population: Two subjects had abnormally low plasma ketorolac concentration-time profiles that were inconsistent with the rest of the elderly population.
Measure: Mean (Standard Deviation); unit: ng*hours/mL
Arm/Group | Ketorolac Tromethamine (Elderly Adults ≥ 65) | Ketorolac Tromethamine (Nonelderly Adults < 65)
Number analyzed (Participants) | 13 | 15
ng*hours/mL | 8794.8 (4129.4) | 6890.8 (3448.5)

5. Primary Outcome: t1/2z (Terminal Half-life)
Time Frame: as for outcome 1
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Ketorolac Tromethamine (Elderly Adults ≥ 65) | Ketorolac Tromethamine (Nonelderly Adults < 65)
Number analyzed (Participants) | 13 | 15
hours | 4.521 (1.142) | 3.313 (0.961)

6. Primary Outcome: MRT (Mean Residence Time)
Time Frame: as for outcome 1
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Ketorolac Tromethamine (Elderly Adults ≥ 65) | Ketorolac Tromethamine (Nonelderly Adults < 65)
Number analyzed (Participants) | 13 | 15
hours | 6.024 (1.496) | 4.441 (1.060)

ADVERSE EVENTS:
Time Frame: 1 month and 1 week
Arm/Group | Ketorolac Tromethamine (Elderly Adults ≥ 65) | Ketorolac Tromethamine (Nonelderly Adults < 65)
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 1/15 | 1/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ketorolac Tromethamine (Elderly Adults ≥ 65) (N=15) | Ketorolac Tromethamine (Nonelderly Adults < 65) (N=15)
Hordeolum (Infections and infestations) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No